CLINICAL TRIAL: NCT02382406
Title: A Phase I/II Study of Carboplatin/Nab-Paclitaxel and Pembrolizumab for Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Carboplatin/Nab-Paclitaxel and Pembrolizumab in NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was completed. It was fully accrued.
Sponsor: Nisha Mohindra, MD (Other)
Collaborators: Hoosier Cancer Research Network (Other); Merck Sharp & Dohme LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Nisha Mohindra, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN13-175
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Results first posted 2022-10-14 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: MK-3475; Pembrolizumab; Carboplatin; Nab-paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; pembrolizumab; Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Phase I Dose Finding Cohort (Experimental): Twelve subjects will be enrolled and treated with carboplatin AUC 6 IV on Day 1, nab-paclitaxel 100 mg/m^2 IV on Day 1, Day 8, and Day 15, pembrolizumab 2* mg/kg IV on Day 1 for 4 cycles. pembrolizumab (Phase I) treatment for Cohort 1 will continue for a maximum duration of 4 21-day cycles
  Phase I, Cohort 1 Maintenance Therapy:
  Participants who have confirmed CR, PR, or SD (non-progression) after 4 cycles, maintenance therapy with MK-3475 2* mg/kg will continue on D1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or a maximum of 2 years from C1D1.
  If unacceptable toxicity is seen in Phase I Cohort 1, 12 additional participants will be enrolled in Cohort 2 and treated with carboplatin AUC 6 IV on D1, nab-paclitaxel 100 mg/m2 IV on D1, D8, and D15, MK-3475 2*mg/kg IV on D1 starting C2. MK-3475 (Phase 1) treatment for Cohort 2 will continue for a maximum duration of 3 21-day cycles (C2-4 only).
  Interventions: Drug: Carboplatin; Drug: Nab-paclitaxel; Drug: MK-3475 (Phase I)
- Arm B: Phase II Investigational Treatment (Experimental): Subjects will be treated with carboplatin AUC 6 given IV on Day 1, nab-paclitaxel 100 mg/m^2 given IV on Day 1, Day 8, and Day 15, and pembrolizumab 200mg IV on Day 1 of each cycle. Pembrolizumab Phase II treatment will continue for a maximum duration of 4 cycles (cycle = 21 days).
  Maintenance Therapy For participants who have confirmed CR, PR, or SD (non-progression) after 4 cycles of induction therapy, maintenance therapy with MK-3475 2* mg/kg will continue on Day 1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or for a maximum of 2 years from C1D1.
  *As additional data from ongoing trials becomes available, the dose of MK-3475 may be adjusted.
  Interventions: Drug: Carboplatin; Drug: Nab-paclitaxel; Drug: MK-3475 (Phase II)

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC 6 IV, D1 for 4 cycles (cycle = 21 days)
  Other Names: Paraplatin
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/m2 IV, D1, D8, D15 for 4 cycles (cycle = 21 days)
  Other Names: Abraxane
Drug: MK-3475 (Phase I) — MK-3475 2 mg/kg IV, D1 for 4 cycles (Cohort 1) or 3 cycles (Cohort 2) (cycle = 21 days)
  Maintenance MK-3475 2 mg/kg IV continues every 21 days after Cycle 4 for up to 2 years.
  Other Names: Pembrolizumab
  Arms: Arm A: Phase I Dose Finding Cohort
Drug: MK-3475 (Phase II) — MK-3475 200 mg IV Day 1 of each cycle (cycle = 21 days)
  Maintenance MK-3475 2 mg/kg IV continues every 21 days after Cycle 4 for up to 2 years.
  Other Names: Pembrolizumab
  Arms: Arm B: Phase II Investigational Treatment

SUMMARY:
This is a phase I/II study for previously untreated subjects with advanced NSCLC. The study will take place in two phases. First, a cohort of twelve participants will be enrolled in phase I part and will be treated with carboplatin, nab-paclitaxel and pembrolizumab. A cohort of twelve subjects will be evaluated for safety and tolerability after 2 cycles of therapy. All subjects who receive either nab-paclitaxel or pembrolizumab will be evaluable. If 33% of subjects or less have unacceptable toxicity in the first cohort or any subsequent cohort (if necessary), the study will proceed to the Phase II part. If more than 33% have unacceptable toxicity, 12 additional subjects will be enrolled in a second cohort, if necessary. If unacceptable toxicity is seen in more than 33% in Cohort 2, the study will end due to unacceptable toxicity of this drug combination.

The phase II part of the study is a single arm study. All subjects will be treated with carboplatin, nab-paclitaxel, and pembrolizumab in 21-day cycles for up to 4 cycles.

Mandatory pre-treatment tumor biopsies will be obtained prior to initiating treatment for all subjects (only if adequate archived samples are unavailable). Mandatory tumor biopsies will be obtained in the Phase II part of the study after 4 cycles of study treatment or at the time of progression, whichever comes first.

For subjects without progression of disease after Cycle 4, pembrolizumab will continue every 3 weeks for up to 2 years or until unacceptable toxicity.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

INVESTIGATIONAL TREATMENT:

Phase I, Cohort 1 Induction Therapy:

* Carboplatin AUC 6 IV, Day 1
* Nab-paclitaxel 100 mg/m^2 IV, Days 1, 8, 15
* pembrolizumab 2 mg/kg IV, Day 1
* Cycle length: 21 days; number of cycles: 4

Phase I, Cohort 1 Maintenance Therapy:

For subjects who have confirmed CR, PR, or SD (non-progression) after 4 cycles of induction therapy, maintenance therapy with pembrolizumab 2* mg/kg will continue on Day 1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or for a maximum of 2 years from Cycle 1, Day 1 (C1D1). Subjects who complete 24 months of treatment with pembrolizumab may be eligible for up to one year of additional study treatment if they progress after stopping study treatment provided they continue to meet inclusion criteria requirements.

If unacceptable toxicity is seen in Phase I, Cohort 1, 12 additional participants will be enrolled.

Phase I, Cohort 2 Induction Therapy (if necessary):

* Carboplatin AUC 6 IV, Day 1
* Nab-paclitaxel 100 mg/m^2 IV, Days 1, 8, 15
* pembrolizumab 2 mg/kg IV, Day 1 (cycle 2-4 only)
* Cycle length: 21 days; Number of cycles: 4

Phase I, Cohort 2 Maintenance Therapy:

For subjects who have confirmed CR, PR, or SD (non-progression) after 4 cycles of induction therapy, maintenance therapy with pembrolizumab 2* mg/kg will continue on Day 1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or for a maximum of 2 years from Cycle 2, Day 1 (C2D1). Subjects who complete 24 months of treatment with pembrolizumab may be eligible for up to one year of additional study treatment if they progress after stopping study treatment provided they continue to meet inclusion criteria requirements.

Phase II Induction Therapy:

* Carboplatin AUC 6 IV, Day 1
* Nab-paclitaxel 100 mg/m^2 IV, Days 1, 8, 15
* pembrolizumab 200mg IV, Day 1 of each cycle
* Cycle length: 21 days; number of cycles: 4

Phase II Maintenance Therapy:

For subjects who have confirmed CR, PR, or SD (non-progression) after 4 cycles of induction therapy, maintenance therapy with pembrolizumab 200 mg will continue on Day 1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or for a maximum of 2 years from Cycle 1, Day 1 (C1D1). Subjects who complete 24 months of treatment with pembrolizumab may be eligible for up to one year of additional study treatment if they progress after stopping study treatment provided they meet the requirements.

*As additional data from ongoing trials becomes available, the dose of pembrolizumab may be adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide written informed consent for the trial and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Subjects must be ≥ 18 years of age.
* Individuals with stage IIIB or IV, unresectable non-small cell lung cancer (NSCLC) who have not received prior chemotherapy for Stage IIIB or IV disease, and who are not candidates for curative surgery or radiation therapy.
* ECOG performance status (PS) 0-1
* Measurable disease by RECIST v1.1 criteria
* Prior to registration, all subjects must have archival tissue available. For subjects who have no archival tissue, but have PD-L1 testing results using the Dako 22C3 antibody, subjects will be permitted to enroll without submitting tissue. If the patient has not had prior testing and no acceptable archival tissue is available, subjects must be willing to consent to providing a pre-treatment biopsy for PD-L1 testing. Regardless of PD-L1 testing status, archival tissue will be requested for research testing if available.
* Phase II subjects must be willing to consent to providing a mandatory post-treatment core biopsy for research if clinical feasible.
* Women are eligible to participate if they are of non-childbearing potential or have documentation of a negative pregnancy test (serum or urine β-hCG) within 3 days of registration. Sexually active pre-menopausal women of childbearing potential must agree to use adequate, highly effective contraceptive measures, starting with the first dose of study drug and for 120 days after the last dose of last study drug. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; (b) oral, implantable, or injectable contraceptives plus one barrier method; or (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥ 1 year.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of last study drug.

Exclusion Criteria:

* Individuals with the presence of symptomatic CNS metastases requiring radiation treatment, surgery, or ongoing use of corticosteroids.
* Untreated or brain metastasis causing any symptoms, such as neurologic deficits or headache. Individuals with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of study drug and any neurologic symptoms have returned to baseline and whole brain radiation or stereotactic radiosurgery completed over 4 weeks prior to registration), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment.
* History of solid organ or stem cell transplant requiring immunosuppressive medications.
* Any prior adjuvant cytotoxic chemotherapy within 12 months of registration. Subjects who received chemotherapy for earlier stage disease more than 12 months prior to study registration are eligible for this trial.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Any radiotherapy within 2 weeks prior to registration (4 weeks for brain radiotherapy as noted above).
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* History of other invasive malignancy that is currently active and/or has been treated within 12 months of registration. (Notable exceptions include: basal cell carcinoma, squamous cell carcinoma of the skin, localized prostate cancer, in situ carcinomas of the cervix and breast, and superficial bladder cancers [non-muscle-invasive]).
* Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Pulmonary conditions such as sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or hypersensitivity pneumonitis.
* Has a history of pneumonitis that required steroids or current pneumonitis.
* Pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE v 4.0 criteria.
* Known significant liver disease including viral, alcoholic, active hepatitis B or C, and/or cirrhosis.
* Abnormal liver or renal function as defined as: bilirubin ≥ 1.5 mg/dL; AST or ALT ≥ 2.5 x the ULN; alkaline phosphatase > 2.5 x the ULN, there is no upper limit if bone metastasis is present in the absence of liver metastasis; creatinine > 1.5 mg/dL
* Abnormal baseline hematologic or coagulation parameters as defined as: absolute neutrophil count (ANC) <1.5 x 10^9/L; hemoglobin < 9.0 g/dL; platelets < 100 x 10^9/L; International Normalized Ratio (INR) of prothrombin time (PT) ≥ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) ≥ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Known activating EGFR mutation or ALK translocation
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Mohindra, M.D., Study Chair — Hoosier Cancer Research Network
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Center, Indianapolis, Indiana
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — https://hoosiercancer.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Cohort 1: Phase I, Cohort 1: Induction Therapy
  Twelve subjects will be enrolled to Cohort 1 and treated with carboplatin AUC 6 IV on Day 1, nab-paclitaxel 100 mg/m^2 given IV on Days 1, 8, and 15, and pembrolizumab 2* mg/kg IV on Day 1.Treatment will continue for a maximum duration of 4 cycles with cycle length of 21 days.
  Phase I, Cohort 1 Maintenance Therapy:
  Participants who have confirmed CR, PR, or SD (non-progression) after 4 cycles, maintenance therapy with pembrolizumab 2* mg/kg will continue on D1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or a maximum of 2 years from C1D1.
- Phase I, Cohort 2: Phase I, Cohort 2: Induction Therapy
  If unacceptable toxicity is seen in Phase I, Cohort 1, 12 additional subjects will be enrolled in Phase I, Cohort 2. Subjects will be treated with carboplatin AUC 6 given IV on Day 1 and nabpaclitaxel 100 mg/m2 given IV on Days 1, 8, and 15. Pembrolizumab 2* mg/kg IV will be given on Day 1 starting in cycle 2. Treatment will continue for a maximum duration of 4 cycles (pembrolizumab given Cycles 2 to 4 only).
  Phase I, Cohort 2 Maintenance Therapy:
  For subjects who have confirmed CR, PR, or SD (non-progression) after 4 cycles of induction therapy, maintenance therapy with pembrolizumab 2* mg/kg will continue on Day 1 of each 21- day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or for a maximum of 2 years from Cycle 2, Day 1.
- Phase II: Induction Therapy Cycles 1-4
  Subjects will be treated with carboplatin AUC 6 given IV on Day 1, nab-paclitaxel 100 mg/m2 given IV on Days 1, 8, and 15, and pembrolizumab 200 mg IV on Day 1. Treatment will continue for a maximum duration of 4 cycles of study treatment. Each cycle starts when all the criteria to start a new cycle are met. A cycle is defined only when you can give all 3 drugs on Day 1, and it coincides with pembrolizumab. Pembrolizumab should be given with carboplatin and nab-paclitaxel on day 1 of the cycle. Chemotherapies may be withheld for six weeks, while pembrolizumab can be withheld for 12-weeks. If there is a pembrolizumab-specific toxicity requiring pembrolizumab to be held, chemotherapy should be resumed without pembrolizumab within 6 weeks if it is felt that chemotherapy is safe by the site investigator. Delays in chemotherapy beyond 6 weeks require withdrawal from the study treatment.
  Maintenance Therapy
  For subjects who have confirmed CR, PR, or SD (non-progression) after 4 cycles of induction therapy, maintenance therapy with pembrolizumab 200 mg will continue on Day 1 of each 21-day cycle. Treatment will continue until progression of disease, unacceptable toxicity, or for a maximum of 2 years from Cycle 1 Day 1.
Period: Study Treatment
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2 | Phase II
Started | 14 | 0 | 32
Completed | 0 | 0 | 2
Not Completed | 14 | 0 | 30
Not completed — Disease Progression | 8 | 0 | 20
Not completed — AE/ Side Effects/ Complications | 4 | 0 | 6
Not completed — Patient withdrawal after therapy start | 1 | 0 | 1
Not completed — symptomatic deterioration | 1 | 0 | 1
Not completed — Death | 0 | 0 | 2
Period: Follow up
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2 | Phase II
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 14 | 0 | 32
Completed | 0 | 0 | 2
Not Completed | 14 | 0 | 30
Not completed — Death | 11 | 0 | 19
Not completed — Symptomatic deterioration | 1 | 0 | 1
Not completed — Patient Refused Follow-up | 1 | 0 | 0
Not completed — Study Terminated | 1 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: No subjects had been enrolled to Phase I, Cohort 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2 | Phase II | Total
Number analyzed (Participants) | 14 | 0 | 32 | 46
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 76] |  | 65.5 [39 to 79] | 65.5 [39 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 |  | 13 | 22
  Male | 5 |  | 19 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 |  | 0 | 0
  Race: Asian | 0 |  | 1 | 1
  Race: Black or African American | 1 |  | 5 | 6
  Race: Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Race: Unknown | 4 |  | 0 | 4
  Race: White | 9 |  | 26 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 |  | 0 | 0
  Ethnicity: Non-Hispanic | 11 |  | 31 | 42
  Ethnicity: Unknown | 3 |  | 1 | 4
Histology Subtype [Count of Participants; unit: Participants]
  Adenocarcinoma | 10 |  | 11 | 21
  Clear Cell (non-component) | 0 |  | 0 | 0
  Clear Cell Component | 0 |  | 0 | 0
  Large Cell Carcinoma | 0 |  | 0 | 0
  Micropapillary Variant | 0 |  | 0 | 0
  Non-Small Cell Lung Cancer, NOS | 0 |  | 1 | 1
  Other | 0 |  | 0 | 0
  Papillary | 0 |  | 0 | 0
  Poorly Differentiated Carcinoma | 0 |  | 3 | 3
  Sarcomatoid | 0 |  | 0 | 0
  Small Cell Carcinoma | 0 |  | 0 | 0
  Squamous Cell Carcinoma | 4 |  | 17 | 21
  Transitional Cell Carcinoma | 0 |  | 0 | 0
Substance use : Number of Cigarettes [Count of Participants; unit: Participants] — The codes are explained as follows :
  1. Never a Smoker
  2. Current Smoker
  3. Former Smoker
  9: Not collected
  Participants
    1 | 2 |  | 1 | 3
    2 | 2 |  | 6 | 8
    3 | 10 |  | 25 | 35
    9 | 0 |  | 0 | 0
Substance use : Number of Cigars [Count of Participants; unit: Participants] — The codes are explained as follows :
  1. Never a Smoker
  2. Current Smoker
  3. Former Smoker
  9: Not collected
  Participants
    1 | 7 |  | 25 | 32
    9 | 7 |  | 7 | 14
Substance use : Number of pipefuls [Count of Participants; unit: Participants] — The codes are explained as follows :
  1. Never a Smoker
  2. Current Smoker
  3. Former Smoker
  9: Not collected
  Participants
    1 | 7 |  | 26 | 33
    9 | 7 |  | 6 | 13
ECOG [Count of Participants; unit: Participants] — ECOG Performance status is explained as :
  0 Fully active; no performance restrictions.
  1 Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  Participants
    0 | 6 |  | 8 | 14
    1 | 8 |  | 23 | 31
    Missing | 0 |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Recommended Phase II Dose
Description: To determine the recommended Phase II dose (RP2D) of MK-3475 and evaluate the safety and tolerability of the combination of MK-3475 with carboplatin/nab-paclitaxel for the first line treatment of phase I participants with advanced NSCLC per CTCAE v4.0 criteria by summarizing the number of adverse events experienced by subjects.
Time Frame: Begin C1D1 and every 2 chemotherapy cycles (6 weeks) thereafter, for up to 2 years or until unacceptable toxicity.
Population: No subjects had been enrolled to Phase I, cohort 2.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I, Cohort 2: Phase I, Cohort 2: Induction Therapy
  If unacceptable toxicity is seen in Phase I, Cohort 1, 12 additional subjects will be enrolled in Phase I, Cohort 2. Subjects will be treated with carboplatin AUC 6 given IV on Day 1 and nabpaclitaxel 100 mg/m2 given IV on Days 1, 8, and 15. Pembrolizumab 2* mg/kg IV will be given on Day 1 starting in cycle 2. Treatment will continue for a maximum duration of 4 cycles (pembrolizumab given Cycles 2 to 4 only).
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2
Number analyzed (Participants) | 14 | 0
Participants
  Patient had at least one adverse event of any grade | 14 | 0
  Patient had at least one grade 3 or greater adverse event | 14 | 0
  Patient had at least one grade 3 or greater treatment related adverse event | 12 | 0
  Patient having serious adverse event | 8 | 0

2. Primary Outcome: Phase II: Disease Assessment for Progression-Free Survival (PFS)
Description: To evaluate progression-free survival (PFS) for phase II participants receiving MK-3475 and carboplatin/nab-paclitaxel for the first line treatment of advanced NSCLC per RECIST 1.1 criteria. PFS is defined as the duration of time from date of registration to time of progression or death, whichever occurs first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of registration to time of first documented progression or death, whichever occurs first (estimate 9 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 32
months | 6.2 [4.6 to 8.5]

3. Primary Outcome: Phase II: Objective Response Rate
Description: To evaluate objective response rate for phase II participants receiving MK-3475 and carboplatin/nab-paclitaxel for the first line treatment of advanced NSCLC per RECIST 1.1 criteria.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the start of treatment until progression or death up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II
Number analyzed (Participants) | 32
Participants | 16

4. Secondary Outcome: Phase I: Disease Assessment for Progression-Free Survival (PFS)
Description: To evaluate progression-free survival (PFS) and objective response for phase I participants receiving MK-3475 and carboplatin/nab-paclitaxel for the first line treatment of advanced NSCLC per RECIST 1.1 criteria.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of registration to time of first documented progression or death, whichever occurs first (estimate 9 months)
Population: No subjects had been enrolled to Phase I, Cohort 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2
Number analyzed (Participants) | 14 | 0
months | 5.2 [4.1 to NA] — upper limit has not been achieved due to insufficient number of participants with events. |

5. Secondary Outcome: Phase I : Objective Response Rate
Description: To evaluate objective response rate for phase II participants receiving MK-3475 and carboplatin/nab-paclitaxel for the first line treatment of advanced NSCLC per RECIST 1.1 criteria.
  Objective response rate (ORR), is defined as the proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: From the start of treatment until progression or death up to 11 months.
Population: No subjects had been enrolled to Phase I, Cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2
Number analyzed (Participants) | 14 | 0
Participants | 1 |

6. Secondary Outcome: Phase I: Disease Assessment for Anti-Tumor Activity
Description: To evaluate anti-tumor activity for phase I participants will be reported as a percentage change in the sum of the dimensions of all measurable lesions as defined by RECIST 1.1 criteria.
Time Frame: From date of registration to time of first documented progression. (Measurable disease will be assessed after every 2 chemotherapy cycles [every 6 weeks thereafter for up to 2 years or until unacceptable toxicity]).
Population: No subjects had been enrolled to Phase I, cohort 2.
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2
Number analyzed (Participants) | 14 | 0
percent change | -6.9457 [-11.3 to 0.578] |

7. Secondary Outcome: Phase I: Overall Survival (OS)
Description: To evaluate overall survival rates for phase I participants receiving MK-3475 and carboplatin/nab-paclitaxel for the first line treatment of advanced NSCLC.
Time Frame: From date of registration to date of death from any cause up to 49 months.
Population: No subjects had been enrolled in Phase I. cohort 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2
Number analyzed (Participants) | 14 | 0
months | 13 [7.1 to 36] |

8. Secondary Outcome: Phase II: Overall Survival (OS)
Description: To evaluate overall survival rates for phase II participants receiving MK-3475 and carboplatin/nab-paclitaxel for the first line treatment of advanced NSCLC.
Time Frame: From date of registration to date of death from any cause up to 42 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 32
months | 16 [12 to NA] — upper limit has not been achieved due to insufficient number of participants with events.

9. Secondary Outcome: Phase II: Disease Assessment for Anti-Tumor Activity
Description: as for outcome 6
Time Frame: as for outcome 6
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Phase II
Number analyzed (Participants) | 32
percent change | -46.7731 [-51.7 to -35.1]

10. Secondary Outcome: Phase II: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To evaluate the safety and tolerability of the combination of MK-3475 with carboplatin/nab-paclitaxel for the first line treatment of phase II participants with advanced NSCLC per CTCAE v4.0. Safety and tolerability is defined as rates of Grade 1-5 toxicity according to CTCAE v4.
Time Frame: Begin C1D1 and every 2 cycles (6 weeks) thereafter, for up to 2 years or until unacceptable toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II
Number analyzed (Participants) | 32
Participants
  Patient had at least one adverse event of any grade. | 32
  Patient had at least one grade 3 or greater adverse event. | 31
  Patient had at least one grade 3 or greater treatment related adverse event. | 27
  Patient having serious adverse event. | 11

11. Secondary Outcome: All Phases: Assessment of Association of PD-L1 Expression on PFS
Description: To evaluate the association of PD-L1 expression on PFS for all participants receiving MK-3475. PD-L1 will be categorized as positive (≥50% expression) or negative (<50% expression) from pre-treatment and post-treatment biopsies. PFS will be summarized by PD-L1 expression.
Time Frame: as for outcome 6
Population: 34 of the 46 subjects have staining information available
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Subjects With PD-L1 Staining Information: PFS was analyzed for 34 patients based on their PD-L1 staining intensity.
Arm/Group | Subjects With PD-L1 Staining Information
Number analyzed (Participants) | 34
months
  >=50% | 4.6 [2.9 to NA] — upper limit has not been achieved due to insufficient number of participants with events.
  0-49% | 4.2 [3.9 to NA] — upper limit has not been achieved due to insufficient number of participants with events.
  0% | 5.6 [3.9 to NA] — upper limit has not been achieved due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Begin C1D1 and every 2 chemotherapy cycles (6 weeks) thereafter, for up to 2 years or until unacceptable toxicity.
Description: No subjects had been enrolled in Phase 1 Cohort 2.
Arm/Group | Phase I, Cohort 1 | Phase I, Cohort 2 | Phase II
All-Cause Mortality (participants affected / at risk) | 11/14 | 0/0 | 19/32
Serious Adverse Events (participants affected / at risk) | 8/14 | 0/0 | 11/32
Other Adverse Events (participants affected / at risk) | 14/14 | 0/0 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Cohort 1 (N=14) | Phase I, Cohort 2 (N=0) | Phase II (N=32)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
INTRA-ABDOMINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CONFUSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
EDEMA LIMBS (General disorders) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ILEAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Cohort 1 (N=14) | Phase I, Cohort 2 (N=0) | Phase II (N=32)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (4) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 4 (7)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 4 (5)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 17 (35)
ANEMIA (Blood and lymphatic system disorders) | 9 (33) | 0 (0) | 19 (58)
ANOREXIA (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 16 (41)
ANXIETY (Psychiatric disorders) | 6 (7) | 0 (0) | 11 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 6 (8)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0) | 5 (8)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0) | 7 (11)
CHEILITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
CHILLS (General disorders) | 1 (1) | 0 (0) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 6 (8) | 0 (0) | 17 (28)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 0 (0) | 14 (23)
CREATININE INCREASED (Investigations) | 3 (5) | 0 (0) | 4 (7)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (3) | 0 (0) | 4 (4)
DIARRHEA (Gastrointestinal disorders) | 4 (14) | 0 (0) | 16 (48)
DIZZINESS (Nervous system disorders) | 3 (3) | 0 (0) | 7 (7)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5)
DYSGEUSIA (Nervous system disorders) | 3 (4) | 0 (0) | 7 (8)
DYSPEPSIA (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 0 (0) | 10 (27)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 2 (2) | 0 (0) | 6 (7)
EDEMA TRUNK (General disorders) | 1 (1) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 7 (7)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 11 (19) | 0 (0) | 29 (88)
FEVER (General disorders) | 3 (3) | 0 (0) | 3 (6)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 2 (4) | 0 (0) | 6 (17)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3) | 0 (0) | 9 (10)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5)
HOT FLASHES (Vascular disorders) | 3 (4) | 0 (0) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (18) | 0 (0) | 3 (5)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
HYPERTENSION (Vascular disorders) | 6 (30) | 0 (0) | 13 (20)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 6 (13)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 11 (24)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 7 (25)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0) | 4 (8)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 0 (0) | 7 (9)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (2) | 0 (0) | 2 (4)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 10 (13)
LOCALIZED EDEMA (General disorders) | 1 (2) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 4 (4)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 4 (13)
MALAISE (General disorders) | 1 (1) | 0 (0) | 2 (2)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (8)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 3 (5)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 8 (13) | 0 (0) | 21 (56)
NECK EDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 12 (32) | 0 (0) | 25 (77)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (3) | 0 (0) | 5 (7)
PAIN (General disorders) | 1 (2) | 0 (0) | 7 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 4 (4)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (3)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 (4) | 0 (0) | 8 (9)
PLATELET COUNT DECREASED (Investigations) | 9 (24) | 0 (0) | 22 (52)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (7)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 12 (28)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (4)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 6 (11)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 7 (8) | 0 (0) | 4 (7)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0) | 4 (6)
THROMBOEMBOLIC EVENT (Vascular disorders) | 3 (3) | 0 (0) | 2 (2)
TRACHEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 6 (10)
VAGINAL INFLAMMATION (Reproductive system and breast disorders) | 1 (4) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 4 (5) | 0 (0) | 10 (22)
WEIGHT LOSS (Investigations) | 3 (8) | 0 (0) | 7 (10)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (5) | 0 (0) | 12 (35)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (3)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
BILIARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BLOATING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
BLURRED VISION (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC TROPONIN I INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 0 (0) | 0 (0) | 4 (4)
CONFUSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 0 (0) | 0 (0) | 5 (7)
FACIAL NERVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 0 (0) | 3 (5)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
GUM INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (15)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (11)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
PAPULOPUSTULAR RASH (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PARESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 2 (5)
PERSONALITY CHANGE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (10)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (6)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
WEIGHT GAIN (Investigations) | 0 (0) | 0 (0) | 2 (3)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT02382406/Prot_SAP_000.pdf